CLINICAL TRIAL: NCT03109496
Title: Study of the Upper Respiratory Tract Microbiota and the Potential of Probiotics for the Treatment of Chronic Otitis Media With Effusion.
Brief Title: The URT and Middle Ear Microbiota in Health and During Chronic OME
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Ethisch Comité, UZA, prof. dr. Olivier Vanderveken, MD, PhD, University Hospital, Antwerp
Other Study IDs: B300201731724
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Otitis Media With Effusion; Healthy
Keywords: OME; Otitis Media with Effusion; Microbiota; Microbiome; URT; Upper Respiratory Tract; Healthy URT microbiota
MeSH Terms: conditions — Otitis Media with Effusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples with extracted DNA (extraction kit targets bacterial DNA) Original samples in glycerol (100 µL) of otitis media patients (for potential future isolation of otitis media associated bacteria)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OME Patients: Suffer from chronic Otitis Media with Effusion (OME) for at least 3 months and undergo ventilation tube placement.
  Interventions: Other: Collection of body fluids/swabs
- Healthy Control: Undergo surgery that gives access to the middle ear space (e.g. cochlear implant surgery) or adenoids, in absence of upper respiratory tract infections.
  Interventions: Other: Collection of body fluids/swabs

INTERVENTIONS:
Other: Collection of body fluids/swabs — Middle ear, ear duct, anterior nare, nasopharynx, adenoids. Niches depend on accessibility for each individual participant.

SUMMARY:
This study analyses which bacteria are present in the middle ear space and adjacent upper respiratory tract niches in healthy people and in patients suffering from chronic otitis media with effusion (OME; glue ear). The aim is to identify and isolate bacteria that are more common and more abundant in healthy people and to evaluate their potential to protect against bacteria commonly involved in OME and other upper respiratory tract infections.

To this end, samples will be collected from both groups (healthy vs OME) and analysed through sequencing of the bacterial 16S gene. In addition, samples obtained from healthy participants will be cultivated to isolate bacteria of interest.

ELIGIBILITY:
Inclusion Criteria:

* Controls: undergo a surgery that gives access to the middle ear space (at least 30 participants; e.g. cochlear implant recipients) or the adenoids.
* OME patients: have fluid accumulation in the middle ear space for 3+ months and receive ventilation tubes. May also undergo adenoidectomy.

Exclusion Criteria:

* Acute upper respiratory tract infections (including acute otitis media)
* Chronic upper respiratory tract infections (except OME in patient group)
* URT malformations (e.g. as seen in people with Down Syndrome or cleft palate)
* Cystic fibrosis
* Autoimmune diseases or immunodeficiency
* Pregnancy
* Use of antibiotics or steroids 1 week before surgery

Ages: 1 Year to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 100 healthy participants vs 100 OME patients.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Microbiota differences between the healthy and diseased URT and middle ear space | Appr. 4 years
  The composition of the bacterial community will be determined through sequencing of the bacterial 16S gene and compared between the participant groups. Species over-represented in healthy participants will be investigated further.

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jorissen J, van den Broek MFL, De Boeck I, Van Beeck W, Wittouck S, Boudewyns A, Van de Heyning P, Topsakal V, Van Rompaey V, Wouters I, Van Heirstraeten L, Van Damme P, Malhotra-Kumar S, Theeten H, Vanderveken OM, Lebeer S. Case-Control Microbiome Study of Chronic Otitis Media with Effusion in Children Points at Streptococcus salivarius as a Pathobiont-Inhibiting Species. mSystems. 2021 Apr 20;6(2):e00056-21. doi: 10.1128/mSystems.00056-21. PMID 33879499